CLINICAL TRIAL: NCT05195151
Title: Modulation of Immune Responses to COVID-19 Vaccination by an Intervention on the Gut Microbiota: a Randomized Controlled Trial
Brief Title: Modification of the COVID-19 Vaccine Response by an Intervention on the Intestinal Flora
Acronym: PIRATES-COV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EG9-179473
Record Dates: First submitted 2022-01-13; First posted 2022-01-18 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: COVID-19; Vaccine Reaction; Elderly
Keywords: Probiotics; COVID-19 Vaccine; Elderly; Immunity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): taking a capsule containing the probiotics 15 d before and 15 d after booster shot.
  Interventions: Dietary Supplement: Taking capsule containing probiotics or placebo
- Control (Placebo Comparator): taking a capsule containing a placebo 15 d before and 15 d after booster shot.
  Interventions: Dietary Supplement: Taking capsule containing probiotics or placebo

INTERVENTIONS:
Dietary Supplement: Taking capsule containing probiotics or placebo — The probiotics capsule containing two strains of probiotics.

SUMMARY:
The elderly, who are often in poorer health, have been particularly affected by the COVID-19 pandemic. Recent study results show that while vaccines have been very effective in the short term, protection for the elderly may not be sufficient 6 months after the 2nd dose. Some countries have started to offer a 3rd dose. We are considering acting on the intestinal flora of the elderly (which is often unbalanced) in order to increase the effectiveness of the vaccination. Indeed, it has been demonstrated that probiotics (which can rebalance the intestinal flora) significantly increase the production of antibodies after vaccination against the flu virus. Our hypothesis is that taking probiotics one month before and one month after the 4th dose of COVID vaccine would result in longer lasting vaccine protection in seniors. This study will include 688 seniors, aged 65-89 years, who have not had COVID-19, who have received 3 doses of an mRNA vaccine and who will accept a another booster dose . All participants will take 1 capsule/day (probiotics or placebo) for 1 month and in the middle of this period will receive a booster dose. On 3 occasions (inclusion, 3 months and 6 months post-vaccination), they will prick their fingertip and express the drop of blood on a blotting paper. They will mail this dried blood sample in an envelope for antibody testing in Quebec Research center. A subgroup of 100 participants willing to travel at CHUS' Clinical Research Center for 2 times (inclusion visit and final visit) will be invited to do a blood test. The investigators expect to reduce the number of seniors who are poorly protected by a booster dose 6 months after the injection. If successful, this approach could quickly be implemented worldwide as probiotics have few side effects and are affordable.

DETAILED DESCRIPTION:
The elderly are at high risk of morbidity and mortality from COVID-19. They are particularly targeted by recent data: i) faster decline of the immune response in the elderly and ii) increase of COVID infection 6 months after the 2nd dose of vaccine. In addition, they often have an imbalance of the microbiota that plays a key role in the activation of the immune system. Taking probiotics, which improve the microbiota, could increase the vaccine response of the elderly. Indeed, it has been shown in 2 meta-analyses that probiotics improve immune response after influenza vaccination. The investigators believe that probiotics taken at the time of 4th dose (booster dose) of vaccine could improve immune memory: i) humoral (cellular Receptor-Binding Domain antibody) and ii) (B lymphocytes, CD4+ T and CD8+ T), in the medium term and would then allow a greater spacing of the booster doses in the future OBJECTIVE: To reduce by 33% the percentage of elders without RBD antibodies, 6 months after the booster dose of vaccine, by taking 2 strains of probiotics compared to placebo. Secondary objectives: To improve the evolution of RBD Ac by longitudinal analysis at 5 different time points (inclusion, vaccination, 1 month, 3 months, and 6 months post-vaccination).- To compare the evolution of neutralizing Ac and memory B, CD4+ T, and CD8+ T cells, at inclusion and 6 months post-vaccination. METHODOLOGYDesign. A randomized, intention-to-treat, blinded, placebo-controlled trial.Investigation products are: for the intervention group, a capsule with 2 strains of probiotics and for control group or a placebo capsule. Participants will take one capsule per day for 30 days (15 d and 15 d after the booster dose of vaccine). Both vaccines (Pfizer-BioNTech, Moderna) may be used depending on availability and state of knowledge . With 1:1 allocation, via the REDCap application, using permuted blocks and stratified according to randomization.gender, age (65-79 and 80-89 years) and vaccine type for the booster dose. Inclusion criteria: (Pfizer-BioNTech or Moderna) for more than 6 months, volunteers for booster dose of vaccine, telephone or internet access, informed consent, and living <75 km from CRC (only for participants for blood test visits). Exclusion criteria: patients with allergies (soy...), COVID-19 disease, possibly affected cognitive functions, chronically weakened immune system (AIDS...) or undergoing anti-cancer treatment. Five finger-prick dried blood samples (DBS) are planned (inclusion, vaccination, 1, 3 and 6 months post-vaccination).The DBS will be mailed to Quebec City . A telephone or mail follow up will be realised for each participant. A subgroup of 100 participants willing to travel will be invited to visit us at the inclusion and final visit to do a blood test. Fecal self-sampling (inclusion) for microbiota study will be sent to I Laforest-Lapointe's laboratory. The levels of RBD Ac and N Ac will be determined by a validated Elisa test (3 time points). From the venous blood samples (inclusion and 6 months post-vaccination),we will be studied: i) the pseudotyped viral neutralization and ii) the cellular immune memory in flow cytometry (B, T CD4+ and T CD8+ lymphocytes). With 30% undetectable RBD Ac in the placebo group (6 months post-vaccine) and 20% in the intervention group, are required (15% attrition, 80% power, 5% two-sided test). The 688 subjects primary analysis on the dichotomous criterion (Ac RBD) will use a GMM logistic regression model for longitudinal data with covariate variant/time.PROJECT OUTCOMEImproving vaccination and spacing vaccine doses among the elderly are major public health issues. If successful, probiotics could be used worldwide very quickly. They have few side effects, are available over the counter and are affordable.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* aged 65-89 years
* who have received 3 doses of a mRNA vaccine (Pfizer-BioNTech or Moderna) for more than 6 months;
* volunteered for a booster dose
* had telephone or internet access
* were able to provide informed consent
* lived <75 km from the CRC (subgroup of 100 participants only)

Exclusion Criteria:

* Patients with COVID-19 disease (clinical and serological data at post);
* with possibly affected cognitive functions (score < 12 on the Functional Activities Questionnaire (FAQ))
* with allergies (soy, lactose, yeast, maltodextrin)
* with a chronically weakened immune system (AIDS...)
* undergoing anti-cancer treatment (chemotherapy or radiotherapy)
* who do not speak French or English.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Male or Female
Enrollment: 592 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Receptor-Binding Domain (RBD) antibodies, 6 months after the vaccine booster shot | inclusion, 3 and 6 months
  The RBD antibody level will be determined by a validated ELISA test (95% sensitivity and 100% specificity). The primary outcome measure is a dichotomous measure of RBD antibodies (detectable or undetectable). The positivity threshold was defined based on the mean optical density (colorimetric reaction on blotting paper) of negative sera +3 SD. Possibly, a quantitative variable will be available.

SECONDARY OUTCOMES:
Anti-N Antibodies | inclusion, 3 and 6 months
  The Anti-N antibodies will be determined by the same procedure than for the dichotomous RBD antibody level (90% sensitivity and 95% specificity).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, Dr, Study Director — Université de Sherbrooke
Locations (1):
- Centre de recherche clinique du CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pasquier JC, Plourde M, Ramanathan S, Chaillet N, Boivin G, Laforest-Lapointe I, Allard-Chamard H, Baron G, Beaulieu JF, Fulop T, Genereux M, Masse B, Robitaille J, Valiquette L, Bilodeau S, H Buch D, Piche A. P robiotics i nfluencing r esponse of a ntibodies over t ime in s eniors after CO VID-19 v accine (PIRATES-COV): a randomised controlled trial protocol. BMJ Open. 2025 Mar 18;15(3):e088231. doi: 10.1136/bmjopen-2024-088231. PMID 40107677

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT05195151/SAP_000.pdf